CLINICAL TRIAL: NCT02982200
Title: The MEDINA Study: Medina Embolization Device In Neurovascular Aneurysms Study - A Post Market Clinical Follow-up Study
Brief Title: Medina Embolization Device In Neurovascular Aneurysm Study
Acronym: MEDINA
Status: Terminated | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: NV-MED-01
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Intracranial Aneurysm
Keywords: Embolization Device; Medina; Rupture Intracranial Aneurysm; Unrupture Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A global prospective, multi-center, single-arm, post-market clinical follow-up (PMCF) study conducted to assess the performance of the Medina Embolization Device when used in unruptured and ruptured intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent using the Ethics Committee-approved consent form and agrees to comply with protocol requirements
* Subject is 18- 85 years old
* Subject has a ruptured or unruptured saccular intra-cranial aneurysm amenable to be treated with the Medina Embolization Device

Exclusion Criteria:

* Aneurysm is partially thrombosed
* Aneurysm has been previously treated with surgery or endovascular therapy
* Subject has had major brain surgery including endovascular procedures within the past 30 days
* Vessel characteristics (tortuosity, stenosis, morphology) preclude safe endovascular access to the aneurysm
* Subject is pregnant or breast-feeding or wishes to become pregnant during the length of the study participation
* The Investigator determines that the validity of the study outcomes may be compromised by the subject's enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Saccular intracranial aneurysm not previously treated.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Complete aneurysm occlusion as defined by the Modified Raymond-Roy Classification (MRRC) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Brouwer, Dr, Study Chair — Karolinska University Hospital
Locations (3):
- Universitätsklinikum Christian Doppler Klinik Salzburg, Salzburg, Austria
- Azienda Ospedaliera Ospedale Niguarda Cà Granda, Milan, Italy
- Hospital Fundación Jiménez Díaz, Madrid, Spain

REFERENCES:
- [Background] Inagawa T, Hirano A. Autopsy study of unruptured incidental intracranial aneurysms. Surg Neurol. 1990 Dec;34(6):361-5. doi: 10.1016/0090-3019(90)90237-j. PMID 2244298
- [Background] Agarwal N, Gala NB, Choudhry OJ, Assina R, Prestigiacomo CJ, Duffis EJ, Gandhi CD. Prevalence of asymptomatic incidental aneurysms: a review of 2,685 computed tomographic angiograms. World Neurosurg. 2014 Dec;82(6):1086-90. doi: 10.1016/j.wneu.2013.01.082. Epub 2013 Jan 19. PMID 23336985
- [Background] Winn HR, Jane JA Sr, Taylor J, Kaiser D, Britz GW. Prevalence of asymptomatic incidental aneurysms: review of 4568 arteriograms. J Neurosurg. 2002 Jan;96(1):43-9. doi: 10.3171/jns.2002.96.1.0043. PMID 11794602
- [Background] Schievink WI. Intracranial aneurysms. N Engl J Med. 1997 Jan 2;336(1):28-40. doi: 10.1056/NEJM199701023360106. No abstract available. PMID 8970938
- [Background] Bonneville F, Sourour N, Biondi A. Intracranial aneurysms: an overview. Neuroimaging Clin N Am. 2006 Aug;16(3):371-82, vii. doi: 10.1016/j.nic.2006.05.001. PMID 16935705
- [Background] Gemmete JJ, Elias AE, Chaudhary N, Pandey AS. Endovascular methods for the treatment of intracranial cerebral aneurysms. Neuroimaging Clin N Am. 2013 Nov;23(4):563-91. doi: 10.1016/j.nic.2013.03.007. Epub 2013 May 25. PMID 24156851
- [Background] Wiebers DO, Whisnant JP, Huston J 3rd, Meissner I, Brown RD Jr, Piepgras DG, Forbes GS, Thielen K, Nichols D, O'Fallon WM, Peacock J, Jaeger L, Kassell NF, Kongable-Beckman GL, Torner JC; International Study of Unruptured Intracranial Aneurysms Investigators. Unruptured intracranial aneurysms: natural history, clinical outcome, and risks of surgical and endovascular treatment. Lancet. 2003 Jul 12;362(9378):103-10. doi: 10.1016/s0140-6736(03)13860-3. PMID 12867109
- [Background] UCAS Japan Investigators; Morita A, Kirino T, Hashi K, Aoki N, Fukuhara S, Hashimoto N, Nakayama T, Sakai M, Teramoto A, Tominari S, Yoshimoto T. The natural course of unruptured cerebral aneurysms in a Japanese cohort. N Engl J Med. 2012 Jun 28;366(26):2474-82. doi: 10.1056/NEJMoa1113260. PMID 22738097
- [Background] Roy D, Milot G, Raymond J. Endovascular treatment of unruptured aneurysms. Stroke. 2001 Sep;32(9):1998-2004. doi: 10.1161/hs0901.095600. PMID 11546888
- [Background] Zuccarello M. Treatment strategy for patients with unruptured intracranial aneurysms. Neurol Med Chir (Tokyo). 2001 Dec;41(12):571-5. doi: 10.2176/nmc.41.571. PMID 11803581
- [Background] Broderick JP, Brott TG, Duldner JE, Tomsick T, Leach A. Initial and recurrent bleeding are the major causes of death following subarachnoid hemorrhage. Stroke. 1994 Jul;25(7):1342-7. doi: 10.1161/01.str.25.7.1342. PMID 8023347
- [Background] Johnston SC, Higashida RT, Barrow DL, Caplan LR, Dion JE, Hademenos G, Hopkins LN, Molyneux A, Rosenwasser RH, Vinuela F, Wilson CB; Committee on Cerebrovascular Imaging of the American Heart Association Council on Cardiovascular Radiology. Recommendations for the endovascular treatment of intracranial aneurysms: a statement for healthcare professionals from the Committee on Cerebrovascular Imaging of the American Heart Association Council on Cardiovascular Radiology. Stroke. 2002 Oct;33(10):2536-44. doi: 10.1161/01.str.0000034708.66191.7d. No abstract available. PMID 12364750
- [Background] Raaymakers TW, Rinkel GJ, Limburg M, Algra A. Mortality and morbidity of surgery for unruptured intracranial aneurysms: a meta-analysis. Stroke. 1998 Aug;29(8):1531-8. doi: 10.1161/01.str.29.8.1531. PMID 9707188
- [Background] Lanzino G, Murad MH, d'Urso PI, Rabinstein AA. Coil embolization versus clipping for ruptured intracranial aneurysms: a meta-analysis of prospective controlled published studies. AJNR Am J Neuroradiol. 2013 Sep;34(9):1764-8. doi: 10.3174/ajnr.A3515. Epub 2013 Apr 11. PMID 23578672
- [Background] Vanninen R, Koivisto T, Saari T, Hernesniemi J, Vapalahti M. Ruptured intracranial aneurysms: acute endovascular treatment with electrolytically detachable coils--a prospective randomized study. Radiology. 1999 May;211(2):325-36. doi: 10.1148/radiology.211.2.r99ap06325. PMID 10228510
- [Background] McDougall CG, Spetzler RF, Zabramski JM, Partovi S, Hills NK, Nakaji P, Albuquerque FC. The Barrow Ruptured Aneurysm Trial. J Neurosurg. 2012 Jan;116(1):135-44. doi: 10.3171/2011.8.JNS101767. Epub 2011 Nov 4. PMID 22054213
- [Background] Molyneux A, Kerr R; International Subarachnoid Aneurysm Trial (ISAT) Collaborative Group; Stratton I, Sandercock P, Clarke M, Shrimpton J, Holman R. International Subarachnoid Aneurysm Trial (ISAT) of neurosurgical clipping versus endovascular coiling in 2143 patients with ruptured intracranial aneurysms: a randomized trial. J Stroke Cerebrovasc Dis. 2002 Nov-Dec;11(6):304-14. doi: 10.1053/jscd.2002.130390. PMID 17903891
- [Background] Seibert B, Tummala RP, Chow R, Faridar A, Mousavi SA, Divani AA. Intracranial aneurysms: review of current treatment options and outcomes. Front Neurol. 2011 Jul 8;2:45. doi: 10.3389/fneur.2011.00045. eCollection 2011. PMID 21779274
- [Background] Im SH, Han MH, Kwon OK, Kwon BJ, Kim SH, Kim JE, Oh CW. Endovascular coil embolization of 435 small asymptomatic unruptured intracranial aneurysms: procedural morbidity and patient outcome. AJNR Am J Neuroradiol. 2009 Jan;30(1):79-84. doi: 10.3174/ajnr.A1290. Epub 2008 Sep 3. PMID 18768715
- [Background] Miller TR, Jindal G, Krejza J, Gandhi D. Impact of Endovascular Technique on Fluoroscopy Usage: Stent-Assisted Coiling versus Flow Diversion for Paraclinoid Internal Carotid Artery Aneurysms. Neuroradiol J. 2014 Dec;27(6):725-31. doi: 10.15274/NRJ-2014-10094. Epub 2014 Dec 1. PMID 25489897
- [Background] Crobeddu E, Lanzino G, Kallmes DF, Cloft HJ. Review of 2 decades of aneurysm-recurrence literature, part 2: Managing recurrence after endovascular coiling. AJNR Am J Neuroradiol. 2013 Mar;34(3):481-5. doi: 10.3174/ajnr.A2958. Epub 2012 Mar 15. PMID 22422182
- [Background] Sekhar LN, Heros RC. Origin, growth, and rupture of saccular aneurysms: a review. Neurosurgery. 1981 Feb;8(2):248-60. doi: 10.1227/00006123-198102000-00020. PMID 7010205
- [Background] Abdihalim M, Watanabe M, Chaudhry SA, Jagadeesan B, Suri MF, Qureshi AI. Are coil compaction and aneurysmal growth two distinct etiologies leading to recurrence following endovascular treatment of intracranial aneurysm? J Neuroimaging. 2014 Mar-Apr;24(2):171-5. doi: 10.1111/j.1552-6569.2012.00786.x. Epub 2013 Jan 14. PMID 23317437
- [Background] Mori K, Nakao Y, Horinaka N, Wada R, Hirano A, Maeda M. Cerebral aneurysm regrowth and coil unraveling after incomplete Guglielmi detachable coil embolization: serial angiographical and histological findings. Neurol Med Chir (Tokyo). 2003 Jun;43(6):293-7. doi: 10.2176/nmc.43.293. PMID 12870547
- [Background] Sedat J, Chau Y, Litrico S, Rasandrarijao D, Lonjon M, Paquis P. Stretched platinum coil during cerebral aneurysm embolization after direct carotid puncture: two case reports. Cardiovasc Intervent Radiol. 2007 Nov-Dec;30(6):1248-51. doi: 10.1007/s00270-007-9058-x. Epub 2007 May 17. PMID 17508233
- [Background] Mascitelli JR, Moyle H, Oermann EK, Polykarpou MF, Patel AA, Doshi AH, Gologorsky Y, Bederson JB, Patel AB. An update to the Raymond-Roy Occlusion Classification of intracranial aneurysms treated with coil embolization. J Neurointerv Surg. 2015 Jul;7(7):496-502. doi: 10.1136/neurintsurg-2014-011258. Epub 2014 Jun 4. PMID 24898735
- [Background] Rouchaud A, Brinjikji W, Gunderson T, Caroff J, Gentric JC, Lanzino G, Cloft HJ, Kallmes DF. Validity of the Meyer Scale for Assessment of Coiled Aneurysms and Aneurysm Recurrence. AJNR Am J Neuroradiol. 2016 May;37(5):844-8. doi: 10.3174/ajnr.A4616. Epub 2015 Nov 12. PMID 26564443
- [Background] McDougall CG, Johnston SC, Gholkar A, Barnwell SL, Vazquez Suarez JC, Masso Romero J, Chaloupka JC, Bonafe A, Wakhloo AK, Tampieri D, Dowd CF, Fox AJ, Imm SJ, Carroll K, Turk AS; MAPS Investigators. Bioactive versus bare platinum coils in the treatment of intracranial aneurysms: the MAPS (Matrix and Platinum Science) trial. AJNR Am J Neuroradiol. 2014 May;35(5):935-42. doi: 10.3174/ajnr.A3857. Epub 2014 Jan 30. PMID 24481333
- [Background] Pierot L, Delcourt C, Bouquigny F, Breidt D, Feuillet B, Lanoix O, Gallas S. Follow-up of intracranial aneurysms selectively treated with coils: Prospective evaluation of contrast-enhanced MR angiography. AJNR Am J Neuroradiol. 2006 Apr;27(4):744-9. PMID 16611757
- [Background] Pierot L, Cognard C, Anxionnat R, Ricolfi F; CLARITY Investigators. Endovascular treatment of ruptured intracranial aneurysms: factors affecting midterm quality anatomic results: analysis in a prospective, multicenter series of patients (CLARITY). AJNR Am J Neuroradiol. 2012 Sep;33(8):1475-80. doi: 10.3174/ajnr.A3003. Epub 2012 Apr 19. PMID 22517279